CLINICAL TRIAL: NCT01522742
Title: Monitoring and Modifying Atherosclerosis in Psoriasis Patients Study
Acronym: MMAPPS
Status: Terminated | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2011P-000557
Record Dates: First submitted 2011-12-29; First posted 2012-02-01 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
Keywords: psoriasis; cardiovascular disease risk; atherosclerosis; etanercept (enbrel)
MeSH Terms: conditions — Psoriasis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy control subjects: Healthy control subjects matched to psoriasis patients on traditional cardiovascular risk factors will be studied at baseline.
- Psoriasis patients starting etanercept: Patients with moderate to severe psoriasis with or without arthritis who are about to be started on etanercept (enbrel) by their treating clinicians will be studied at baseline and 3 months after etanercept therapy.

SUMMARY:
The main aims of this study are to determine whether: a) psoriasis patients with or without arthritis have more cardiovascular inflammation than healthy subjects and b)3 months of etanercept (enbrel) therapy (prescribed to psoriasis patients with or without arthritis by their treating clinicians) will decrease cardiovascular inflammation.

DETAILED DESCRIPTION:
Psoriasis is a common disease characterized by skin lesions and systemic inflammation with or without arthritis. Patients with psoriasis have a higher risk of cardiovascular disease than healthy subjects, and this may be related in part to the inflammatory nature of their disease. This study is intended to help provide explanations for the increased cardiovascular disease risk in psoriasis and to assess whether this risk can be reduced by biologic anti-inflammatory therapies prescribed to resolve skin lesions and arthritis.

ELIGIBILITY:
FOR PSORIASIS PATIENTS

Inclusion Criteria:

-men and women age 18-80 with moderate-to-severe psoriasis (with or without arthritis) newly initiating biologic therapy with etanercept (enbrel) 50 mg once or twice weekly

Exclusion Criteria:

* pregnancy or breastfeeding
* women of child-bearing potential refusing to practice abstinence or to use a reliable barrier form of birth control including condoms, IUD, or diaphragm
* history of acute coronary syndrome or coronary artery stenting or surgery, or significant autoimmune/inflammatory disease other than psoriasis or a related psoriatic condition
* previous therapy for psoriasis with a biologic agent within the past 4 months
* new initiation of a statin or antihyperglycemic agent within the past 3 months
* screening hemoglobin < 11
* conditions which would make MDCT coronary angiography/ cardiac FDG-PET protocol unsafe or unfeasible including: significant renal dysfunction with an eGFR by Cockcroft-Gault equation of <60 ml/min, contrast dye allergy, contraindication to beta-blockers (e.g. severe asthma, hypotension, or heart block), or contraindication to nitroglycerin (uninterruptable administration of phosphodiesterase inhibitors), body weight greater than 320 lbs (PET scanner table limitation)
* report by subject of any significant radiation exposure over the course of the year prior to enrollment; significant exposure is defined as:

  * more than 2 myocardial perfusion studies within the past 12 months
  * more than 2 CT angiograms within the past 12 months
* concurrent enrollment in a clinical trial judged by the investigator to introduce concerns about safety or confounding

FOR HEALTHY CONTROL SUBJECTS

Inclusion Criteria:

-men and women age 18-80 without psoriasis

Exclusion Criteria:

* pregnancy or breastfeeding
* women of child-bearing potential refusing to practice abstinence or to use a reliable barrier form of birth control including condoms, IUD, or diaphragm
* history of acute coronary syndrome or coronary artery stenting or surgery, or significant autoimmune/inflammatory disease
* screening hemoglobin < 11
* conditions which would make MDCT coronary angiography/ cardiac FDG-PET protocol unsafe or unfeasible including: significant renal dysfunction with an estimated creatinine clearance by Cockcroft-Gault equation of <60 ml/min, contrast dye allergy, contraindication to beta-blockers (e.g. severe asthma, hypotension, or heart block), or contraindication to nitroglycerin (e.g. continuous administration of phosphodiesterase inhibitors), body weight greater than 320 lbs PET scanner table limitation)
* report by subject of any significant radiation exposure over the course of the year prior to enrollment; significant exposure is defined as:

  * more than 2 myocardial perfusion studies within the past 12 months
  * more than 2 CT angiograms within the past 12 months
* concurrent enrollment in a clinical trial judged by the investigator to introduce concerns about safety or confounding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with moderate-to-severe psoriasis with or without arthritis will be recruited primarily from dermatology and rheumatology clinics in the eastern Massachusetts area.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Aortic/coronary target to background ratio (TBR) on cardiac FDG-PET. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Degree of aortic/coronary atherosclerotic plaque inflammation assessed via cardiac FDG-PET as target to background ratio (TBR) of the standardized uptake value (SUV).

SECONDARY OUTCOMES:
Aortic/coronary atherosclerotic plaque burden on MDCT coronary angiography. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Burden of aortic/coronary atherosclerotic plaque as measured by MDCT coronary angiography.
Aortic/coronary atherosclerotic plaque morphology on MDCT coronary angiography. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Morphology of the aortic/coronary atherosclerotic plaque (e.g. calcification score, vulnerability characteristics) as measured by MDCT coronary angiography.
Endothelial function as measured by flow-mediated vasodilation. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
Oral glucose tolerance. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Blood sugar and insulin levels during a standard 2-hour oral glucose tolerance test.
Lipid and lipoprotein levels. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Levels of total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, apolipoprotein A1, apolipoprotein B, apolipoprotein C-II, apolipoprotein C-III, and apolipoprotein E.
Inflammatory biomarker levels. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Levels of inflammatory biomarkers including but not limited to high-sensitivity C-reactive protein, interleukin-6, and TNF-alpha.
Body fat distribution. | Baseline in all subjects and change from baseline to 3 months in psoriasis cohort starting etanercept (enbrel).
  Measurements of height, weight, waist-to-hip ratio, leg circumference, arm circumference, and neck circumference. Determinations by whole body DEXA scanning of the total body and regional percent fat and lean body mass. Determination by single-slice abdominal computed tomography of total fat area, visceral adipose tissue, and subcutaneous adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States